CLINICAL TRIAL: NCT02047357
Title: Participatory Intervention to Reduce Maternal Depression and Under Five Child Morbidity- A Cluster-Randomized Controlled Trial
Brief Title: Participatory Intervention to Reduce Maternal Depression and Under Five Child Morbidity
Acronym: ROSHNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Grand Challenges Canada (Other); The Hincks-Dellcrest Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ROS-PILL-001; LTP-PLUS 001 (Other Grant/Funding Number: Grand Challenges Canada)
Record Dates: First submitted 2014-01-21; First posted 2014-01-28 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Maternal Depression
Keywords: Maternal depression; Mother; Child; LTP; Learning Through Play; Healthy thinking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Experimental): Learning Through Play Plus
  Interventions: Other: Learning Through Play Plus
- Control (No Intervention): This arm will receive no intervention

INTERVENTIONS:
Other: Learning Through Play Plus — Learning Through Play (LTP) Plus is a low-literacy, sustainable program intended to provide parents with information on the healthy growth and development of their young children. The LTP research-based activities enhance children's development while simultaneously promoting attachment security through building parents' ability to read and be sensitive to their children's cues and through active involvement in their children's development. Plus the Thinking Healthy Program (THP) which adopts 'here and now' problem-solving approach. THP uses cognitive behavior therapy (CBT) techniques of active listening, changing negative thinking, and collaboration with the family.
  Other Names: Psycho social intervention
  Arms: Intervention Arm

SUMMARY:
To test the efficacy of an innovative affordable intervention program that can be used by non-specialists, including mothers and lady health workers with minimal training in low resource countries such as Pakistan

DETAILED DESCRIPTION:
Specific challenges: In Pakistan rates of depression particularly in women are high, as well as other risks to the growth and development of young children and child mortality. Numerous studies provide compelling evidence that maternal depression not only affects mothers but is also associated with long term emotional, cognitive and behavioural problems in children. Depressed mothers are unable to provide primary care necessary for growth of their children during the first 3-years of life, a critical period for child development. Disability due to depressive symptoms (such as fatigue, poor concentration, loss of interest) is likely to affect child-care abilities directly, while impaired social functioning is likely to have indirect consequences through lack of support in childcare. Disturbances in mother-infant relationship in depressed mothers negatively influence the child's development. There is now evidence from some low income countries that effectively delivered participatory group interventions are cost effective intervention for improving maternal and child health. The Community-Based participatory Intervention LTP Plus has been designed to address maternal depression and a parenting program of child psychosocial development through mother-infant play providing stimulation, and support for exploration and autonomy for the infant.The proposed study will test the efficacy of an innovative affordable intervention program that can be used by non-specialists, including mothers and lay health workers with minimal training in low resource countries such as Pakistan.

Project Impact: LTP Plus is proposed as a low cost intervention to improve maternal mental and physical health, reduce infant and children under five years' morbidity and mortality, and promote healthy child development. Learning Through Play (LTP) Plus is a low-literacy, sustainable program intended to provide parents with information on the healthy growth and development of their young children. The LTP research-based activities enhance children's development while simultaneously promoting attachment security through building parents' ability to read and be sensitive to their children's cues and through active involvement in their children's development. Plus the Thinking Healthy Program (THP) which adopts 'here and now' problem-solving approach, THP uses cognitive behavior therapy (CBT) techniques of active listening, changing negative thinking, and collaboration with the family.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included in the study if they are:

  * 18 to 44 years old Mothers with children aged between 0-30 months
  * Resident in the trial site catchments area
  * Ability to complete a baseline assessment

Exclusion Criteria:

* Participants will be excluded from the study if they have:

  * A medical disorder that would prevent participation in clinical trial.
  * Temporary resident unlikely to be available for follow up.
  * Active suicidal ideation or any other severe or physical mental disorder

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 774 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
EPDS | Change from Baseline to 3 month
  The EPDS is a self-report questionnaire composed of ten items scored on a four-point scale (0-3) designed to assess pregnancy and postpartum depression Cox et al. (1987).

SECONDARY OUTCOMES:
Knowledge of Expectation and Child Development | Baseline, 3 months and 6 months
  A 20-item questionnaire will be used to assess maternal knowledge and expectations for child development in the first three years. A change in mothers' knowledge was reported for Pakistani mothers who participated in LTP (Rahman et al, 2009).
Patient Health Questionnaire (PHQ) (Kroenke, Spitzer, Williams et al, 2001) | Baseline, 3 month and 6 month
  The Patient health Questionnaire (PHQ) is a simple 10 item self-report questionnaire can also be administered by a trained research worker. A score of 10 or more is taken as cut -off for depressive disorder
Generalized Anxiety Disorder (GAD) 7 (Spitzer, R. L., Kroenke, K., Williams, J. B., & Lowe, B. 2006) | Baseline, 3 month and 6 month
  The GAD-7 is a 7 item scale used to screen for and measure severity of Genralised Anxiety Disorder. Scores of 5, 10 & 15 are taken as cut-off points for mild, moderate and high
Clinical Interview Schedule Revised (CISR) | Baseline, 3 month and 6 month
  The clinical Interview Schedule-Revised is a fully structured diagnostic instrument that was developed from an existing instrument, the Clinical Interview Schedule (CIS), assessing minor psychiatric morbidity in the community, general hospital, occupational and primary care research
Quality of life (EQ 5 D) | Baseline, 3 month and 6 month
  It is a measure of health and quality of life. This is a standardised instrument for use as a measure of health outcome; it provides a simple descriptive profile and a single index value for health status.

OTHER OUTCOMES:
Cost effectiveness analysis | Baseline, 3 month and 6 month
  It is used for evaluating cost effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Batool Fatima, Principal Investigator — Pakistan Institute of Living and Learning; Nancy Cohen, Ph.D, Principal Investigator — The Hincks-Dellcrest Centre
Locations (1):
- Community, Gadap, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Ashraf T, Alvi MH, Ullah A, Kiran T, Gumber A, Sikander S, Chaudhry N, Chaudhry IB, Husain N. Economic evaluation of Learning Through Play Plus in comparison to usual care for depressed mothers alongside a randomised controlled trial. BMC Health Serv Res. 2026 Feb 4. doi: 10.1186/s12913-026-14113-0. Online ahead of print. PMID 41639802
- See also: Pakistan Institute of learning and living — http://pill.org.pk